CLINICAL TRIAL: NCT01596855
Title: A Phase 2, Randomized, Open-Label Active-Comparator (Epoetin Alfa) Dose-Ranging Safety and Exploratory Efficacy Study of FG-4592 in Subjects With End-Stage Renal Disease Receiving Maintenance Hemodialysis (HD)
Brief Title: Study of FG-4592 in Subjects With End-Stage Renal Disease Receiving Maintenance Hemodialysis in China
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Collaborators: Ruijin Hospital (Other); RenJi Hospital (Other); Chang Zheng Hospital (Unknown); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Peking University First Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); First Affiliated Hospital of Zhejiang University (Other); Peking Union Medical College Hospital (Other); Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-4592-048
Record Dates: First submitted 2012-04-30; First posted 2012-05-11 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Anemia in End Stage Renal Disease
Keywords: Anemia; Renal
MeSH Terms: conditions — Anemia | interventions — roxadustat; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FG-4592 (Experimental): Active Drug
  Interventions: Drug: FG-4592
- Epoetin alfa (Active Comparator): Standard of care
  Interventions: Drug: Epoetin Alfa

INTERVENTIONS:
Drug: FG-4592 — TIW dosing, capsule
  Arms: FG-4592
Drug: Epoetin Alfa — TIW
  Arms: Epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of FG-4592 in maintaining and/or correcting hemoglobin (Hb) given to subjects with End Stage Renal Disease (ESRD) on maintenance hemodialysis and receiving epoetin alfa.

DETAILED DESCRIPTION:
Dose ranging study with three consecutive dose escalation cohorts. The study objectives are to demonstrate that FG-4592 is effective in maintaining hemoglobin (Hb) levels when converting from epoetin alfa and to establish optimum starting doses and dose adjustment regimens for Hb maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has voluntarily signed and dated an informed consent form
2. Age 18 to 75 years
3. End-stage renal disease (ESRD) and receiving maintenance hemodialysis TIW for ≥4 months prior to Day 1
4. Hemoglobin (Hb) values in 4 screening visits and the mean Hb must be between 9.0 and 12.0 g/dL (inclusive), and the difference between them must be ≤1.5 g/dL.
5. Stable doses of IV or Subcutaneous injection of epoetin alfa, defined as follows:

   * Epoetin alfa dose range for 6 weeks prior to Day -7:

     3000 to 20,000 IU/week
   * Stable doses of epoetin alfa (i.e., the maximum epoetin alfa dose does not exceed 130% of the lowest dose of epoetin alfa taken in this period)
6. Complete Blood Count (CBC), Hematology, liver function blood tests within acceptable limits
7. Serum folate and vitamin B12 levels above the lower limit of normal (LLN)
8. Body weight: 40 to 100 kg (dry weight) inclusive
9. Body mass index (BMI): 16 to 38 kg/m2 inclusive
10. HD subjects: dialysis vascular access via native arteriovenous fistula or synthetic graft (not via catheter)

Exclusion Criteria:

1. Anticipated change in hemodialysis prescription or access during the screening or dosing period of the study
2. Any clinically significant infection or evidence of an underlying infection such as a white blood cell count (WBC) > ULN during screening on two separate occasions,
3. Positive for any of the following: human immunodeficiency virus (HIV); hepatitis B surface antigen (HBsAg); anti-hepatitis C virus antibody (anti-HCV Ab)
4. History of chronic liver disease
5. New York Heart Association Class III or IV congestive heart failure
6. Chronic inflammatory disease other than glomerulonephritis that could impact erythropoiesis (e.g., systemic lupus erythematosis, rheumatoid arthritis, celiac disease) even if it is currently in remission
7. Active or chronic gastrointestinal bleeding, or a known coagulation disorder
8. Hemoglobinopathy (e.g., homozygous sickle-cell disease, thalassemia of all types, etc.)
9. Hematological disorders, including myelodysplastic syndrome, multiple myeloma, or pure red cell aplasia
10. History of hemosiderosis, hemochromatosis, polycystic kidney disease, or anephric
11. Active hemolysis or diagnosis of hemolytic syndrome
12. Known bone marrow fibrosis
13. Uncontrolled or symptomatic secondary hyperparathyroidism (PTH>600ng/L)
14. Any prior organ transplantation
15. Drug-treated gastroparesis, short-bowel syndrome, or any other gastrointestinal condition that may lead to reduced absorption of study drug
16. History of alcohol or drug abuse; or a positive drug screen for a substance that has not been prescribed for the subject
17. Prior treatment with FG-4592
18. Use of traditional Chinese medicines (TCM) during the screening visit to Day 1 or plans to use TCM during the study unless approved in advance by the Medical Monitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin maintenance using FG-4592 dosing regimen in ESRD subjects. Number of subjects who hemoglobin levels are maintained at no lower than 0.5 g/dL below their mean baseline value during weeks 6 and 7. | Week 7

SECONDARY OUTCOMES:
Number (%) of subjects whose hemoglobin levels are between 9.0 and 13.0 g/dL at Weeks 3, 4, 5, 6 and 7. | Week 7
Number (%) of subjects whose hemoglobin levels at Weeks 3, 4, 5, 6 and 7 are greater than or equal to their baseline level. | Week 7

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - First Affiliated Hospital, Sun Yat-Sen University, Guangzhou
  - Zhejiang University No 1. Hospital, Hangzhou
  - Chang Zheng Hospital, Shanghai
  - Renji Hospital, Shanghai
  - RuiJin Hospital, Shanghai
  - XinHua Hospital, Shanghai
  - ShenZhen People's Hospital, Shenzhen

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278